CLINICAL TRIAL: NCT00424502
Title: An Open-label Study to Evaluate the Effect of MabThera on Treatment Response in Patients With Rheumatoid Arthritis Who Have Had an Inadequate Response to Previous TNF Inhibition.
Brief Title: A Study of MabThera (Rituximab) in Patients With Rheumatoid Arthritis Who Have Had an Inadequate Response to a TNF-Blocker.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML20538
Record Dates: First submitted 2007-01-18; First posted 2007-01-19 (Estimated); Results first posted 2014-07-14 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab; Methotrexate

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: rituximab [MabThera/Rituxan]; Drug: Methotrexate

INTERVENTIONS:
Drug: rituximab [MabThera/Rituxan] — 1g iv on days 1 and 15
  Other Names: MabThera/Rituxan
Drug: Methotrexate — 10-25mg po/week

SUMMARY:
This single arm study will evaluate the efficacy and safety of MabThera in patients with active rheumatoid arthritis whose current treatment with one or more TNF blocker had produced an inadequate response. Patients will receive MabThera (1g infusion) on day 1 and day 15, and will continue on their basic methotrexate therapy (10-25mg/week). The anticipated time on study treatment is 3-12 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* diagnosed RA for >=3 months prior to first administration of study medication;
* inadequate response or intolerance to >=1 anti-TNF therapies, alone or in combination with methotrexate;
* if using NSAIDS, analgesics or oral corticosteroids, must be on a stable dose for >=2 weeks prior to start of study.

Exclusion Criteria:

* other chronic inflammatory diseases;
* use of parental corticosteroids within 4 weeks prior to screening;
* severe heart failure, or severe, uncontrolled cardiac disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-01; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- Hungary (2):
  - Budapest
  - Debrecen

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab 1000 Milligrams (mg): Participants received rituximab 1000 mg intravenously (IV) and methylprednisolone 100 mg IV on Days 0 and 14.
Period: Overall Study
Arm/Group | Rituximab 1000 Milligrams (mg)
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Rituximab 1000 mg: Participants received rituximab 1000 mg IV and methylprednisolone 100 mg IV on Days 0 and 14.
Arm/Group | Rituximab 1000 mg
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.70 (12.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Disease Activity Score Based on 28-Joint Count (DAS28)
Description: DAS28 consists of swollen joint count (SJC) and tender joint count (TJC) measurements, erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hr]), and Patient Global Assessment of Disease Activity (participant-rated assessment of arthritis) with transformed scores ranging from 0 to 10. Higher scores indicated greater affectation due to disease activity. DAS28 equal to or less than (≤)3.2 equals (=) low disease activity, greater than (>)3.2 to 5.1 = moderate to high disease activity.
Time Frame: Day 0 and Week 24
Population: All enrolled participants who received at least one dose of study treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rituximab 1000 mg
Number analyzed (Participants) | 20
units on a scale
  Day 0 | 6.03 (0.96)
  Week 24 | 4.01 (1.49)
Statistical Analysis 1: Comparison: Rituximab 1000 mg; Change from Baseline to Week 24; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 2.017, 95% CI 2-sided [1.39 to 2.64], Standard Deviation 1.34

2. Secondary Outcome: Health Assessment Questionnaire - Disability Index (HAQ-DI) Scores
Description: The HAQ-DI score consists of questions referring to 8 categories: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and common daily activities. For each of the categories, participants reported the amount of difficulty they had in performing 2 or 3 specific subcategory items. The standard disability score was calculated from the 8 categories by dividing the sum of the individual categories by the number of categories answered, yielding a score from 0 (without any difficulty) to 3 (unable to do).
Time Frame: Day 0 and Week 24
Population: All enrolled participants. n (number) = number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rituximab 1000 mg
Number analyzed (Participants) | 20
units on a scale
  Day 0 (n=20) | 1.14 (0.31)
  Week 24 (n=19) | 0.87 (0.36)
Statistical Analysis 1: Comparison: Rituximab 1000 mg; Change from baseline to Week 24; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 0.276, 95% CI 2-sided [0.151 to 0.401], Standard Deviation 0.259

3. Secondary Outcome: Anti-cyclic Citrullinated Peptide (Anti-CCP)
Description: Anti-CCP measured as absorbance units per milliliter (AU/mL).
Time Frame: Day 0 and Week 24
Population: All participants who received at least 1 dose of study drug; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: AU/mL
Arm/Group | Rituximab 1000 mg
Number analyzed (Participants) | 20
AU/mL
  Day 0 (n=20) | 731.07 (569.83)
  Week 24 (n=19) | 846.41 (988.18)

4. Secondary Outcome: Vascular Endothelial Growth Factor (VEGF)
Description: VEGF was measured as picograms per milliliter (pg/mL).
Time Frame: Day 0 and Week 24
Population: All participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Rituximab 1000 mg
Number analyzed (Participants) | 20
pg/mL
  Day 0 | 516.68 (523.89)
  Week 24 | 520.15 (451.10)

5. Secondary Outcome: Erythrocyte Sedimentation Rate (ESR)
Description: ESR was measured in mm/hr.
Time Frame: Day 0 and Week 24
Population: All participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Rituximab 1000 mg
Number analyzed (Participants) | 20
mm/hr
  Day 0 | 45.25 (22.40)
  Week 24 | 30.85 (4.58)
Statistical Analysis 1: Comparison: Rituximab 1000 mg; Change from baseline to Week 24; Test type: Superiority or Other; p = 0.012, t-test, 2 sided; Mean Difference (Final Values) = 14.40, 95% CI 2-sided [3.52 to 25.28], Standard Deviation 23.24

6. Secondary Outcome: C-Reactive Protein (CRP)
Description: CRP was measured in milligrams per liter (mg/L).
Time Frame: Day 0 and Week 24
Population: All participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Rituximab 1000 mg
Number analyzed (Participants) | 20
mg/L
  Day 0 | 6.13 (9.77)
  Week 24 | 4.32 (6.51)
Statistical Analysis 1: Comparison: Rituximab 1000 mg; Change from baseline to Week 24; Test type: Superiority or Other; p = 0.337, t-test, 2 sided; Mean Difference (Final Values) = 1.81, 95% CI 2-sided [-2.03 to 5.65], Standard Deviation 8.21

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and serious AEs (SAEs) were reported up to Week 48.
Arm/Group | Rituximab 1000 mg
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 9/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab 1000 mg (N=20)
Mood change (Psychiatric disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Blood in stool (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Throat pain (Gastrointestinal disorders) | 2
Fever (General disorders) | 2
Dry eye sensation (Eye disorders) | 1
Blurred vision (Eye disorders) | 1
Feeling of weakness (General disorders) | 1
Sleep disturbance (Psychiatric disorders) | 1
Leucopenia (Blood and lymphatic system disorders) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Progression of rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1
Haemorrhagic suffusion (Blood and lymphatic system disorders) | 1
Acute conjunctivitis (Eye disorders) | 1
Infusion site pruritus (Injury, poisoning and procedural complications) | 1
Infusion site swelling (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.